CLINICAL TRIAL: NCT02964299
Title: Mandibular Advancement Bite Block Efficacy Observational Study
Status: Completed | Type: Observational
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-04-003C
Record Dates: First submitted 2016-10-26; First posted 2016-11-16 (Estimated); Last update posted 2016-11-16 (Estimated); Status verified 2016-11

CONDITIONS: Airway Obstruction
Keywords: Gastrointestinal endoscopy; Moderate sedation; Airway management
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard: Standard bite block
- Mandibular advancement bite block: Mandibular advancement by 3 mm, 6 mm or 9 mm from neutral position
  Interventions: Device: Mandibular advancement bite block

INTERVENTIONS:
Device: Mandibular advancement bite block — Mandibular advancement bite block that provides mandibular advancement by 3 mm, 6 mm, or 9 mm from neutral position
  Groups: Mandibular advancement bite block

SUMMARY:
The purpose of this study is to compare the effect of mandibular advancement bite block to standard bite block for prevention of hypoxemia, intervention events and adverse effects during endoscopic examinations.

DETAILED DESCRIPTION:
During endoscopic examinations, especially upper gastrointestinal, bile duct, or bronchoscopic examinations, the endoscope need to be placed through the mouth. A bite block is used to protect vulnerable endoscope and protect patient's teeth. During sedative endoscopic exams, respiratory depression, apnea or upper airway obstruction will occur under the influence of the sedative medications. Serious adverse events may occur such as hypoxemia. A nasal airway, Larson's maneuver, jaw thrust or chin lift may be needed to open airways.

Mandibular advancement devices has been widely used in treating obstructive sleep apnea. A modified bite block that provides mandibular advancement could provide entry inlet of endoscope as well as provide mandibular advancement to provide patent airway during sedative endoscopy. In this study, we group the patients into test group using mandibular advancement bite block and a control group using standard bite block. After anesthetic induction, gastric endoscopy was performed. Degree of upper airway obstruction will be evaluated and recorded. Differences between the two groups will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist class I or II
* Patients undergoing routine upper gastrointestinal endoscopy under sedation

Exclusion Criteria:

* Baseline oxygen saturation < 90%
* Known difficult airway
* Oral or facial surgery history
* BMI > 35
* patients with gastroparesis or gastrointestinal bleeding
* anticipated exam time > 30 minutes

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ASA class I or II patients admitted for routine upper gastrointestinal endoscopy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Area under curve of 95% oxygen desaturation | up to 30 minutes
  From start of sedation drug administration to end of endoscopic examination with the endoscope withdrawal from patient's mouth, peripheral oxygen saturation recorded. Area under curve of 95% oxygen desaturation is calculated by (95-saturation) x time.

SECONDARY OUTCOMES:
number of rescue interventions: chin lift, jaw thrust, insertion of nasal airway or mask-bag ventilation | up to 30 minutes
  From start of sedation drug administration to end of endoscopic examination with the endoscope withdrawal from patient's mouth, number of events such as chin lift, jaw thrust, insertion of nasal airway, or mask-bag ventilation recorded.
Adverse events: partial or complete airway obstruction, or apnea | up to 30 minutes
  From start of sedation drug administration to end of endoscopic examination with the endoscope withdrawal from patient's mouth, number of events such as snoring, stridor, apnea, airway obstruction or loss of end tidal carbon dioxide waveform recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Nung Teng, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Department of Anesthesiology, Taipei Veterans General Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided